CLINICAL TRIAL: NCT04680416
Title: A Tissue Collection Study in Patients With Renal Clear Cell Carcinoma Who Respond to Immune Checkpoint Inhibitors to Identify Targets of Tumor-Reactive T Cells
Brief Title: Tissue Collection to ID TCRs From Renal Clear Cell Carcinoma Patients Responding to Immune Checkpoint Inhibitors
Status: Withdrawn | Type: Observational
Why Stopped: Lack of patient samples
Sponsor: TScan Therapeutics, Inc. (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202005006
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-12

CONDITIONS: Renal Clear Cell Carcinoma
Keywords: Renal Clear Cell Carcinoma; T Cell Receptor-engineered T-cell therapy; Tissue Collection
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
T Cell Receptor-engineered T-cell therapy (TCR T-cell therapy) offers a potentially transformative approach to treating cancer, but is currently limited by the lack of known targets (Maus and June, 2016; Ping et al., 2018). Arguably the most clinically meaningful way to discover new targets and TCRs for TCR T-cell therapy is to study the tumorinfiltrating lymphocytes of patients that are actively responding to immune checkpoint inhibitor (ICI) therapy. These T cells are clonally expanded as a result of checkpoint inhibition and are responsible for the patient's clinical response. The goal of this study is to acquire tumor and blood samples from up to 40 patients with renal cell carcinoma (RCC) malignancies who respond to ICI therapy. T cells will be isolated from these samples and the targets of their TCRs determined using TScan's genome-wide, high-throughput target ID technology. The expected outcome of this study is the discovery of a collection of new targets for TCR T-cell therapy, along with associated TCRs that will then be developed as novel therapies for patients with similar malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Known or suspected diagnosis of renal clear cell carcinoma.
2. Age ≥18 years at time of diagnosis.
3. ECOG performance status 0-2.
4. Ability to understand and willingness to sign an informed consent document.
5. Patients must be eligible for or currently receiving treatment with immune checkpoint inhibitor (ICI) therapy as determined by the patient's treating oncologist. The treatment regimen may comprise more than one agent but must include at least one ICI drug.

   Examples of FDA-approved ICI drugs include pembrolizumab (Keytruda), nivolumab (Opdivo), atezolizumab (Tecentriq), avelumab (Bavencio), durvalumab (Imfinzi), cemiplimab (Libtayo), and ipilimumab (Yervoy). Immune-checkpoint inhibitors not on this list may also be used, provided they are FDA-approved.
6. Patients undergoing an on-treatment biopsy must show a partial response of one or more lesions, as assessed by the investigator, using RECIST 1.1 or irRECIST criteria.
7. Patients undergoing surgical resection of residual tumors must show a partial response by RECIST 1.1 or irRECIST criteria of at least one of the resected lesions.
8. Patients undergoing an on-treatment biopsy must have a cancer lesion that is amenable for biopsy under local anesthesia or moderate sedation per standard procedures. The tumor biopsy must have an acceptable clinical risk, as judged by the investigator.
9. Platelet count ≥50×109 /L prior to biopsy or per the service performing the biopsy.
10. Absolute neutrophil count ≥1500×103 /L.
11. Must be able to safely hold aspirin, clopidogrel (Plavix), prasugrel (Effient), cangrelor (Kengreal), or ticagrelor (Brilinta) for ≥5 days prior to biopsy.
12. Not receiving therapeutic anticoagulation at the time of the biopsy. Patients on therapeutic anticoagulation must be able to safely hold anticoagulation for the procedure with an acceptable risk, as judged by the investigator. Patients who are on anticoagulation for clinical reasons and deemed appropriate for biopsy must be OFF anticoagulation prior to biopsy as follows:

    1. No warfarin (Coumadin) for 5 days.
    2. No low-molecular weight heparin (LMWH; e.g. dalteparin/ Fragmin, enoxaparin/ Lovenox) for 24 hours.
    3. No fondaparinux/ Arixtra for 48 hours.
    4. Patients receiving alternative forms of anticoagulation not listed above (e.g., dabigatran, rivaroxaban, apixaban, edoxaban) should consult with the prescribing physician and the service performing the biopsy regarding safety and administration guidelines prior to biopsy. Bleeding risks with these agents should be considered when deciding on whether to perform the biopsy if for research purposes only.

Exclusion Criteria:

1. Concurrent disease or condition that would make the patient inappropriate for study participation, or any serious medical or psychiatric disorder that would interfere with the subject's safety.
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
3. History of serious or life-threatening allergic reaction to local anesthetics (i.e., lidocaine, xylocaine).
4. Pregnant women are excluded because there may be an increased risk to both mother and fetus in the setting of moderate sedation, which is required for biopsies of certain anatomic sites (e.g., liver, lung, bone). Also, ionizing radiation from CT-guided biopsies may pose a risk to the unborn fetus.
5. Active cardiac disease, defined as:

   * Uncontrolled or symptomatic angina within the past 3 months.
   * History of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes). Atrial fibrillation with controlled ventricular response on treatment is not an exclusion.
   * Myocardial infarction < 6 months from study entry.
   * Uncontrolled or symptomatic congestive heart failure.
6. Any other condition, which in the opinion of the patient's treating oncologist or the physician performing the biopsy procedure, would make participation in this protocol unreasonably hazardous for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women and members of all races and ethnic groups are eligible for this protocol. It is expected that the mix of patients entering this study will reflect the demographics of the clinic population seen at the Washington University hospitals and associated clinics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Single Cell Sequencing | 1 year
  Number of patients, through single-cell sequencing, displaying the TCR repertoire of these tumor and blood samples with new targets

CONTACTS AND LOCATIONS:
Overall Officials: James Hsieh, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No